CLINICAL TRIAL: NCT05467657
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation of the Somatosensory Cortex on Motor Learning
Brief Title: Transcranial Magnetic Stimulation on Somtosensory Cortex Enhances Motor Learning in People With Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuron, Spain (Other)
Collaborators: Centro Superior de Estudios Universitarios La Salle (Unknown)
Responsible Party: Principal Investigator, Alfredo Lerín Calvo, Physical Therapist, Neuron, Spain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALC001NR001
Record Dates: First submitted 2021-10-04; First posted 2022-07-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Transcranial Magnetic Stimulation; Stroke; Motor Learning
Keywords: Transcranial magnetic stimulation; Stroke; Motor learning; Somatosensory cortex; Motor function
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The experimental group will recive conventional therapy and repetitive transcranial magnetic stimulation over somatosensory cortex, and control group will receive conventional therapy and sham repetitive transcranial stimulation
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repetitive transcranial magnetic stimulation (Experimental): Participants in the experimental group will receive one hour of rehabilitation therapy daily with 30 minutes of Task Oriented Training (TOT) and 30 minutes of Robotic-Assisted Therapy (RAT), 5 days per week, and repetitive Transcranial Magnetic Stimulation (rTMS) will be applied. This process will comprise 5 weekly sessions of excitatory stimulation over the primary somatosensory area of the participant's affected side. For this purpose, the motor area will be localised and a coil will be placed 2 cm posterior to it. An isolated pulse will be applied to the motor area to ensure that the coil is not placed over the motor area using 110% of the motor resting threshold. After this, 24 trains of 5 Hz at an intensity of 90% of the motor resting threshold will be applied for 10 seconds, with a rest between series of 5 seconds (a total of 1200 pulses).
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): The control group treatment will consist of a daily one-hour session of 30 minutes of task-oriented training (TOT) and 30 minutes of robotic-assisted therapy (RAT), for 5 days per week, to which the repetitive Transcranial Magnetic Stimulation (rTMS) placebo treatment will be added. To achieve the placebo, the localisation of the area to be stimulated will be carried out but the coil will be placed in a vertical position so the current wil not go through the skull and the patient will just feel the vibration, communicating to the participant that it is likely that during the stimulation process he/she will not feel anything.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — It will be applyed a magnetic field over the Somatosensory cortex of the patient that pretends to hiperexcite the membrans of the neurons inthis area to enhance motor learning

SUMMARY:
The purpose of this study is to know the efficacy about the application of repetitive transcranial magnetic stimulation (rTMS) on the somatosensory cortex (S1) to enhance motor function in people with stroke.

DETAILED DESCRIPTION:
Subjects will attend the Neuron rehabilitation clinic or La Beata Hospital on their own to begin a rehabilitation program. After being recruited for the study and signing informed consent an electroencephalography test (EEG) will be performed to determine the absence of ectopic foci and to reduce risks during the treatment process with repetitive transcranial magnetic stimulation (rTMS).

One assessor will be in charge of carrying out the rest of the neurophysiological tests, so the Resting Motor Treshold (RMT) will be collected. To finalise the assessment, a second evaluator will test sensory aspects with the two-point discrimination test, the Semmes-Wenstein monofilaments, the pinprick test and the sterognosia test, and motor aspects by means of the ARAT test.

Once the assessment is completed, the participant will be assigned to the control or experimental group through a randomisation process carried out by another person in the research group using GraphPad software. The control group treatment will consist of a daily one-hour session of 30 minutes of task-oriented training (TOT) and 30 minutes of robotic-assisted therapy (RAT), for 5 days per week, to which the rTMS placebo treatment will be added. To achieve the placebo, the localisation of the area to be stimulated will be carried out but the coil will be placed in a vertical position so the current wil not go through the skull and the patient will just feel the vibration, communicating to the participant that it is likely that during the stimulation process he/she will not feel anything.

Participants in the experimental group will receive one hour of rehabilitation therapy daily with 30 minutes of TOT and 30 minutes of RAT, 5 days per week, and rTMS will be applied. This process will comprise 5 weekly sessions of excitatory stimulation over the primary somatosensory area of the participant's affected side. For this purpose, the motor area will be localised and a coil will be placed 2 cm posterior to it. An isolated pulse will be applied to the stimulation area to ensure that the coil is not placed over the motor area using 110% of the motor resting threshold. After this, 24 trains of 5 Hz at an intensity of 90% of the motor resting threshold will be applied for 10 seconds, with a rest between series of 5 seconds (a total of 1200 pulses).

Finally, once the treatment period is over, after 20 sessions, the assessment will be carried out again, recording the initial tests in the same order by the same assessors.

A descriptive analysis of the demographic characteristics and the main and secondary variables in the sample will be performed, presenting the continuous variables as Mean ± Standard Deviation (SD), 95% Confidence Interval (CI), while the categorical variables will be presented as Number (n) and Percentage (relative frequency, %). To measure normality, the Kolmogorov-Smirnov test will be used, and if the quantitative variables show a non-normal distribution, they will be described with the median and the interquartile range. Parametric tests (normal distribution) will be chosen for comparison between groups based on the central limit theorem, in case the sample exceeds 30 subjects per group. Therefore, the mixed-model ANOVA test will be used to analyze the group factor in quantitative variables and the chi-square test for qualitative variables to observe the variability of the intra-group treatment response. In case ANOVA reveals statistical significance, a post-hoc analysis with Bonferroni correction will be performed. A P-value < 0.05 will be accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered an ischaemic or haemorrhagic stroke with more than 3 months of evolution
* Presenting a score >21 points on the Mini-mental State Examination scale.

Exclusion Criteria:

* Severe impairment of upper limb motor function (<15 points on the Fugl-Meyer Assessment Upper Extremity scale)
* Any contraindications to rTMS, such as metal implants, history of epileptic seizures or taking medication that lowers the seizure threshold
* Previous history of neurological pathology.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in electroencephalographic activity | Change from Baseline in electroencephalographic activity at 4 weeks
  The electrical signal evoked by the motor cortex when realizing a movement. It will be measured with an electroencephalograph

SECONDARY OUTCOMES:
Changes in Resting Motor Treshold | Change from Baseline in Resting Motor Treshold at 4 weeks
  Electrophysilogic response of the motor cortex after a sensory stimulation. By placing the stimulator coil over the subject's motor cortex, an electrical pulse is passed to activate the upper motor neurons, generating a motor response that is recorded by electromyography in the subject's interosseous musculature. In this way, the excitability of the corticospinal tract can be measured by observing the latency recorded by electromyography.
Changes in Motor learning | Change from Baseline in Motor learning at 4 weeks
  Ability to learn or demonstrate the ability to acquire, maintain, modify and control voluntary postures and movement patterns with a goal framed motor behaviour.One way to measure this in neurologically affected subjects is through motor dexterity, as it is a variable derived from motor learning that is more useful in the clinical setting. Because of this, Action Research Arm Test (ARAT) will be used. This test asses the motor dexterity of the patient by 4 subtest based on functional movements (grasping, holding, clamping and gross movement)
Changes in Sensitivity | Change from Baseline in Sensitivity at 4 weeks
  It refers to the integration of information received by sensory receptors. It will be measured by the 2 points discrimination test, the Semmes-Weinstein monofilaments and the pinprick test, all of them applyed on tenar eminence of the subject. using an esthesiometer
Changes in Esterognosia | Change from Baseline in esterognosia at 4 weeks
  It refers to the three-dimensional perception and recognition of an object through active touch. To assess sterognosia, the patient, with eyes closed, must recognise a set of objects presented randomly from the ulnar side of the hand and between the fingers and thumb. The objects used for the test are a pencil, a paper clip, a safety pin, a coin, a button, a pill, a rubber band, a string, a spoon, a bucket and a marble, andthe protocol by Van Heest, House and Putnam, 1993 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Lerín Calvo, PhD student, Principal Investigator — Neuron, Spain
Locations (2):
- Spain (2):
  - Neuron Chamberí, Madrid
  - Neuron Madrid Rio, Madrid

IPD SHARING:
Plan to Share IPD: No